CLINICAL TRIAL: NCT03633604
Title: An Expanded IND Access Investigation of HBOC-201 Infusion in Patients With Severe Acute Anemia Who Are Unable to Receive Red Blood Cell Transfusion
Brief Title: Expanded Access IND Administration of HBOC-201 in Patients With Severe Acute Anemia
Status: Available | Type: Expanded Access
Sponsor: Jonathan H. Waters (Other)
Collaborators: HbO2 Therapeutics LLC (Industry)
Responsible Party: Sponsor-Investigator, Jonathan H. Waters, Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Other Study IDs: STUDY19070376
Record Dates: First submitted 2018-08-08; First posted 2018-08-16 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Anemia Severe
Keywords: Hematologic Diseases; Blood Substitutes
MeSH Terms: conditions — Hematologic Diseases | interventions — HBOC 201

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Biological: HBOC-201 — Intravenous administration of a hemoglobin based oxygen carrier (HBOC) in patients with life-threatening anemia, for whom allogeneic blood transfusion is not an option.
  Other Names: Hemopure; hemoglobin glutamer - 250 (bovine)

SUMMARY:
HBOC-201 provides an oxygen treatment bridge and can be used to eliminate, delay, or reduce the need for red blood cell transfusions in anemic patients

This is an expanded access IND protocol, and will provide treatment with HBOC-201 to severely anemic adults for whom blood is not an option

DETAILED DESCRIPTION:
HBOC 201 [hemoglobin glutamer - 250 (bovine)] is an investigational agent, manufactured by Hemoglobin Oxygen Therapeutics LLC (HbO2 Therapeutics), located in Souderton, PA. HBOC-201, has been previously studied17-20 as an alternative to blood transfusions in severely anemic patients needing a way to enhance tissue oxygenation. HBOC-201 is purified, cross-linked and polymerized acellular bovine hemoglobin (Hb) in a modified lactated Ringer's solution, and does not require blood compatibility.

HBOC-201 is an oxygen carrying fluid that increases plasma and total hemoglobin concentration. HBOC-201 has a right-shifted oxygen binding equilibrium curve with a P50 of 40 ± 6 mmHg compared to 27 mmHg for corpuscular hemoglobin. When fully saturated, HBOC-201 binds approximately 1.39 mL of oxygen per gram hemoglobin and, therefore, has the same oxygen carrying capacity as whole blood having the same hemoglobin concentration. To the extent that HBOC-201 administration increases the total hemoglobin concentration in circulation, HBOC-201 is capable of increasing convective oxygen delivery (DO2), defined as the product of blood oxygen content (ml O2/ml blood) and volumetric blood flow (ml blood/min.) At concentrations corresponding to at least 10% of the total hemoglobin concentration, HBOC-201 also facilitates diffusive oxygen delivery, primarily by shortening diffusion distances between RBCs and between RBCs and the endothelium. The higher P50 of HBOC-201 compared to that of cellular hemoglobin further facilitates diffusion of oxygen from RBCs to tissues through increased oxygen off-loading.

HBOC-201 provides an oxygen treatment bridge and can be used to eliminate, delay, or reduce the need for red blood cell transfusions in anemic patients

This is an expanded access IND protocol, and will provide treatment with HBOC-201 to severely anemic adults for whom blood is not an option.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥ 18 years of age
2. Critically ill patients with hemoglobin ≤ 6 g/dL (or 7-8 g/dL with significant active bleeding), and physiologic evidence of critical ischemia, for example: elevated troponins, altered mental status, acute renal failure, lactic acidosis or evidence of central nervous system acute deficits
3. Patients or their Legally Authorized Representative who are able and willing to provide informed consent
4. Blood is not an option due to:

   * refusal of transfusion
   * lack of compatible red blood cells

Exclusion Criteria:

1. Patients with known hypersensitivity or allergy to beef products
2. Patients with pre-existing uncontrolled hypertension, heart failure, renal failure (caution should be exercised if renal insufficiency is present), circulatory hypervolemia or systemic mastocytosis*
3. Patients who are eligible for blood transfusions
4. Patients who are > 80 years old*
5. Pregnant or lactating women

   * on a case by case and quality of life determination

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States